CLINICAL TRIAL: NCT03950440
Title: Assessing the Incidence of Postoperative Delirium Following Aortic Valve Surgery
Brief Title: Assessing the Incidence of Postoperative Delirium Following Aortic Valve Replacement
Acronym: IPOD-AV
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, dr. Danny Hoogma, Anesthesiologist, Universitaire Ziekenhuizen KU Leuven
Other Study IDs: S61710
Record Dates: First submitted 2019-05-08; First posted 2019-05-15 (Actual); Results first posted 2023-02-16 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2022-05

CONDITIONS: Postoperative Delirium; Aortic Valve Stenosis
Keywords: Transaortic valve replacement; Surgical aortic valve replacement; TAVR; SAVR
MeSH Terms: conditions — Emergence Delirium; Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — presence of neural injury markers
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Our primary aim in this observational study is to identify the incidence of POD in the first five postoperative days by using the 3-minute Diagnostic confusion assessment method (3D-CAM), the derived version for intensive care unit (CAM-ICU) or nurse reports in patients undergoing different techniques of aortic valve replacement. Patients are followed 5 days postoperative with the 3D-CAM or until resolution of POD. Six months postoperatively, a follow-up by phone is planned for activity of daily living (ADL).

DETAILED DESCRIPTION:
A significant and often underrecognized complication after surgery is postoperative delirium (POD) causing increased morbidity and mortality. This is especially true for the older cardiac surgical patient, in whom the incidence of POD is up to 70%. Surgical invasiveness and herewith related inflammation, a cholinergic load of medications, postoperative pain or use of opioids are examples of precipitating factors that can be altered to reduce the incidence of POD. Transaortic valve replacement (TAVR) is a revolutionary technique that has led to a dramatic decrease in surgical invasiveness and improved outcomes in high-risk surgical patients. However, only a few studies evaluated neurocognitive outcome after surgical aortic valve replacement (SAVR) compared to TAVR, suggesting a reduced incidence of POD with TAVR compared to SAVR. In contrast, other studies found almost no difference in POD in the aforementioned patient groups. Hence, it remains still unclear which technique best to use in patients at high risk for POD.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to undergo elective

  * TAVI
  * SAVR (with or without coronary artery bypass grafting (CABG) or pulmonary vein isolation (PVI))
* Patient able to read and understand the research materials

Exclusion Criteria:

* Inability to give informed consent
* Presence of delirium at baseline as screened with the 3-minute Diagnostic Confusion Assessment Method (3D-CAM)
* Combined surgical procedures (e.g. mitral valve surgery, aortic surgery or other)

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Any patient presenting for the indicated surgery in a tertiary university hospital
Sampling Method: Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2018-09-23 (Actual); Primary Completion 2020-01-20 (Actual); Study Completion 2020-07-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Danny Hoogma, MD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- University Hospitals Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hoogma DF, Venmans E, Al Tmimi L, Tournoy J, Verbrugghe P, Jacobs S, Fieuws S, Milisen K, Adriaenssens T, Dubois C, Rex S. Postoperative delirium and quality of life after transcatheter and surgical aortic valve replacement: A prospective observational study. J Thorac Cardiovasc Surg. 2023 Jul;166(1):156-166.e6. doi: 10.1016/j.jtcvs.2021.11.023. Epub 2021 Nov 17. PMID 34876283

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Between September 2018 and January 2020, 250 patients were included: 84 patients in the TAVI group and 166 in the SAVR group. During the screening, 43 patients were non eligible (age <70 years, additional valve surgery, already participated or were intubated) and 41 patients were excluded (did not speak Dutch, baseline delirium, declined to participated).
Groups:
- TAVI Patients (n=84): Patients aged ≥ 70 years and scheduled for aortic valve replacement surgery by TAVI
- Mini-sternotomy (n=82): Patients aged ≥ 70 years and scheduled for aortic valve replacement surgery SAVR without concomitant revascularization or surgical ablation for atrial fibrillation thru mini-sternotomy
- Full-sternotomy (n=84): Patients aged ≥ 70 years and scheduled for aortic valve replacement surgery SAVR with or without concomitant revascularization and/or surgical ablation for atrial fibrillation thru full-sternotomy
Period: Overall Study
Arm/Group | TAVI Patients (n=84) | Mini-sternotomy (n=82) | Full-sternotomy (n=84)
Started | 84 | 82 | 84
Primary Analysis | 84 | 82 | 84
1 Month Follow-up | 80 | 82 | 84
Completed (6 month follow-up) | 76 | 80 | 83
Not Completed | 8 | 2 | 1
Not completed — Death | 8 | 2 | 1

BASELINE CHARACTERISTICS:
Population: Baseline characteristics without propensity weighting.
Groups:
- Total: Total of all reporting groups
Arm/Group | TAVI Patients (n=84) | Mini-sternotomy (n=82) | Full-sternotomy (n=84) | Total
Number analyzed (Participants) | 84 | 82 | 84 | 250
Age, Continuous [Mean (Standard Deviation); unit: years] | 83 (5.9) | 78 (5.3) | 78 (5.3) | 80 (5.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 37 | 33 | 102
  Male | 52 | 45 | 51 | 148
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0 | 0
  Unknown or Not Reported | 84 | 82 | 84 | 250
EuroSCORE II [Mean (Standard Deviation); unit: %] | 7.28 (5.98) | 2.47 (1.47) | 5.03 (4.09) | 4.95 (4.68)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Postoperative Delirium
Description: Using the 3-minute Diagnostic confusion assessment method (3D-CAM), the derived version for intensive care unit (CAM-ICU) and nurse reports combined with interview with the caregivers and patient
Time Frame: Until the fifth postoperative day in hospital (an average of 5 days). In case of POD, followup was continued until resolution of POD or discharge (whichever comes first) up to 19 days.
Population: Propensity weighted analysis
Measure: Count of Participants; unit: Participants
Arm/Group | TAVI Patients (n=84) | Mini-sternotomy (n=82) | Full-sternotomy (n=84)
Number analyzed (Participants) | 84 | 82 | 84
Participants | 13 | 41 | 45
Statistical Analysis 1: Comparison: TAVI Patients (n=84) vs Mini-sternotomy (n=82) vs Full-sternotomy (n=84); Frailty scores (Tilburg and essential) and Euroscore were specified in the protocol. Age was added during the meeting before start of the data-analysis; Test type: Other — Propensity scores were obtained from three separate multivariable logistic regression models contrasting each group versus the two other groups. The result from this multivariable model quantifies the degree of separation between both groups; p < 0.0001, Poisson regression — The double robust approach refers to the weighted analysis with all variables involved in the construction of the propensity-based weights added as confounders in the model; Risk Ratio (RR) = 0.26, 95% CI 2-sided [0.16 to 0.44] — TAVI-group compared to the SAVR-group; The double robust approach refers to the weighted analysis with all variables involved in the construction of the propensity-based weights added as confounders in the model

2. Secondary Outcome: Onset Moment of Postoperative Delirium
Description: Moment of onset of POD during the first five postoperative days or until discharge
Time Frame: During the first five postoperative days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | TAVI Patients (n=84) | Mini-sternotomy (n=82) | Full-sternotomy (n=84)
Number analyzed (Participants) | 84 | 82 | 84
days | 4 [2.5 to 4.5] | 3 [2.5 to 5] | 4 [3 to 5]

3. Secondary Outcome: Duration of POD
Description: Duration of delirium in days using the 3D-CAM or ICU-CAM
Time Frame: If POD develops during the first 5 postoperative days, patient will be followed until POD has resolved or until discharge
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | TAVI Patients (n=84) | Mini-sternotomy (n=82) | Full-sternotomy (n=84)
Number analyzed (Participants) | 84 | 82 | 84
days | 4 [2.5 to 8] | 3 [2.5 to 5] | 4 [3 to 6]

4. Secondary Outcome: Severity of POD
Description: assessed with the delirium long severity measure-based confusion assessment method (CAM-S Long). Ten features are evaluated and scored. The first item is either 0 (not present) or 1 (yes). The other 9 features are scored as 0 (not present), 1 (present but mild) or 2 (present and marked). These subscores are than combined on a scale ranging from 0 (no delirium) to 19 (severe delirium).
Time Frame: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | TAVI Patients (n=84) | Mini-sternotomy (n=82) | Full-sternotomy (n=84)
Number analyzed (Participants) | 84 | 82 | 84
score on a scale | 6 [4 to 12] | 5 [3 to 7] | 5 [3 to 7]

5. Secondary Outcome: Number of Patients With Adverse Events According to the Composite Endpoint Early Safety According to VARC-2 at 30 Days
Description: Count of patient having an adverse event according to the composite endpoint "Early safety (at 30 days)" defined by the Valve Academic Research Consortium (VARC)-2. These include: all-cause mortality, all stroke, life threatening bleeding, acute kidney injury stage 2 or 3 and major vascular complications.
Time Frame: Until 30 days postoperatively
Population: Propensity weighted analysis
Measure: Count of Participants; unit: Participants
Arm/Group | TAVI Patients (n=84) | Mini-sternotomy (n=82) | Full-sternotomy (n=84)
Number analyzed (Participants) | 84 | 82 | 84
Participants | 31 | 22 | 20

6. Secondary Outcome: Number of Patients With Adverse Events According to the Composite Endpoint Clinical Efficacy According to VARC-2 at 6 Months
Description: Count of patient having an adverse event according to the composite endpoint "Clinical efficacy (at 6 months)" defined by the Valve Academic Research Consortium (VARC)-2. These include: all-cause mortality, all stroke, rehospitalization, NYHA Classe 3 or 4 and valve dysfunction.
Time Frame: 6 months
Population: Propensity weighted analysis
Measure: Count of Participants; unit: Participants
Arm/Group | TAVI Patients (n=84) | Mini-sternotomy (n=82) | Full-sternotomy (n=84)
Number analyzed (Participants) | 84 | 82 | 84
Participants | 32 | 21 | 18

7. Secondary Outcome: Assessment of Instrumental Activities of Daily Living During 6-months Interview
Description: Assessment of Instrumental activities of daily living (IADL) divided over 7 items. Each item can be scored with either 0 (not capable), 1 (capable with aid) or 2 (without aid). These subscores are summed on a scale ranging from 0 (worse outcome) to 14 (best outcome).
Time Frame: 6 months postoperatively
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TAVI Patients (n=84) | Mini-sternotomy (n=82) | Full-sternotomy (n=84)
Number analyzed (Participants) | 63 | 70 | 66
score on a scale | 8.3 (3.5) | 10.8 (3.2) | 11.1 (3.2)

8. Secondary Outcome: Intensive Care Unit (ICU) Length of Stay
Description: Intensive care unit (ICU) length of stay following the procedure
Time Frame: Until 30 days postoperatively
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | TAVI Patients (n=84) | Mini-sternotomy (n=82) | Full-sternotomy (n=84)
Number analyzed (Participants) | 84 | 82 | 84
hours | 29 [25 to 68] | 47 [26 to 102] | 46 [27 to 76]

9. Secondary Outcome: Hospital Length of Stay
Description: Amount of days hospitalized in the primary center
Time Frame: Until 30 days postoperatively
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | TAVI Patients (n=84) | Mini-sternotomy (n=82) | Full-sternotomy (n=84)
Number analyzed (Participants) | 84 | 82 | 84
days | 4 [3 to 10] | 8 [7 to 12] | 10 [7.5 to 13]

10. Secondary Outcome: Count of Patients Discharged Directly Home
Description: Discharge destination directly after discharge from the hospital back home
Time Frame: Until 30 days postoperatively
Measure: Count of Participants; unit: Participants
Arm/Group | TAVI Patients (n=84) | Mini-sternotomy (n=82) | Full-sternotomy (n=84)
Number analyzed (Participants) | 84 | 82 | 84
Participants | 71 | 47 | 55

ADVERSE EVENTS:
Time Frame: 6 months postoperatively patients were contacted by phone and by mail. Furthermore the general practitioner and/or treating cardiologist was contacted for relevant information.
Arm/Group | TAVI Patients (n=84) | Mini-sternotomy (n=82) | Full-sternotomy (n=84)
All-Cause Mortality (participants affected / at risk) | 8/84 | 2/82 | 1/84
Serious Adverse Events (participants affected / at risk) | 36/84 | 21/82 | 17/84
Other Adverse Events (participants affected / at risk) | 28/84 | 18/82 | 18/84
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TAVI Patients (n=84) (N=84) | Mini-sternotomy (n=82) (N=82) | Full-sternotomy (n=84) (N=84)
All stroke (Nervous system disorders) | 9 (9) | 3 (3) | 3 (3) — According to VARC-2 criteria
Rehospitalization (General disorders) | 9 (9) | 7 (7) | 10 (10)
NYHA 3/44 (Cardiac disorders) | 11 (11) | 8 (8) | 8 (8) — According to VARC-2 criteria
Valve dysfunction (Cardiac disorders) | 13 (13) | 4 (4) | 2 (2) — According to VARC-2 criteria
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TAVI Patients (n=84) (N=84) | Mini-sternotomy (n=82) (N=82) | Full-sternotomy (n=84) (N=84)
Early safety at 30 days (General disorders) | 28 (28) | 18 (18) | 18 (18) — According to VARC-2 criteria

LIMITATIONS AND CAVEATS:
We would like to refer to the published manuscript

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-13): https://cdn.clinicaltrials.gov/large-docs/40/NCT03950440/Prot_SAP_000.pdf